CLINICAL TRIAL: NCT03632057
Title: Shock Efficacy, a Randomized Study Comparing Fixed Tilt and Fixed Pulse Width in a General Implantable-Cardioverter Population
Brief Title: Shock Efficacy Study Comparing Fixed Tilt and Fixed Pulse Width in a General Implantable-Cardioverter Population
Acronym: EFICAZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRD_914
Record Dates: First submitted 2018-07-19; First posted 2018-08-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Ventricular Arrythmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed Tilt (65%) (Active Comparator): This is the control group, so device programming for shock energy is the default setting
  Interventions: Device: Fixed Tilt (65%)
- Fixed Pulse Width (Active Comparator): This is the Study group.
  Interventions: Device: Fixed Pulse Width

INTERVENTIONS:
Device: Fixed Tilt (65%) — This is the standard group, so device programming for shock energy is the default setting
  Arms: Fixed Tilt (65%)
Device: Fixed Pulse Width — The device has to be programmed with fixed pulse width for each phase of the biphasic waveform
  Arms: Fixed Pulse Width

SUMMARY:
This is a prospective, 1:1 randomized, interventional, multicenter and international trial. Approximately 790 subjects are expected to be enrolled to 40 sites in the south of Europe and Middle East.

DETAILED DESCRIPTION:
The objective of this study is to evaluate and compare the efficacy of the first appropriate shock of an ICD in a ventricular tachyarrhythmia, when the waveform of the shock is programmed with the standard waveform, Fixed Tilt with a value of 65% (Control Group), versus the exclusive waveform programmable in SJM ICDs, Fixed Pulse Width (Study Group), in a standard population of subjects with ICD indication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the current ESC indications for ICD or CRT-D implant. This includes upgrades indications from pacemaker to ICD or to CRT-D or replacements of ICDs or CRT-Ds provided that there is no previous record of ineffective shocks

  * Subjects who are willing to be registered on the Merlin.net remote follow-up program
  * Subject ≥18 years
  * Subjects with life expectancy of at least 1 year
  * Subjects who agree to comply with the follow-up program included in this protocol

Exclusion Criteria:

* • Subjects on the waiting list for a heart transplant or under consideration for a transplant over the next 12 months

  * Subjects with Myocardial infarction or unstable angina within 40 days prior to enrollment
  * Subjects who have undergone a recent cardiac revascularization (PTCA, Stent or CABG) procedure in the 4 weeks prior to enrollment
  * Functional NYHA Class IV
  * Subjects who are participating in another ICD or CRT-D study
  * Subjects who are pregnant at the time of enrollment or women of childbearing potential that do not take contraceptives
  * Any disability or limitations to correctly understand or complete the study (physical, intellectual, logistical)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of the first appropriate shock to revert a tachyarrhythmia to sinus rhythm | 5 years
  Rate of rhythm conversion from Ventricular Tachyarrhythmia to sinus rhythm by the first appropriate shock programmed to 25 Joules (or equivalent voltage) programming the shock waveform in Fixed Pulse Width (Study Group) versus the Fixed Tilt with value 65% (Control Group).

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Fernandez, MD, Principal Investigator; Javier Alzueta, MD, Principal Investigator
Locations (2):
- Spain (2):
  - Hospital Virgen de la Victoria, Málaga, Andalusia
  - Hospital Puerta de Hierro, Madrid

IPD SHARING:
Plan to Share IPD: No